CLINICAL TRIAL: NCT04513392
Title: Comparison of Treatment Outcome of Blue Light Laser and KTP Laser for Benign Vocal Fold Lesions: A Randomized Trial
Brief Title: Comparison of BL and KTP Laser for Treatment of Benign Vocal Fold Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, R. Jun Lin, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v1.0
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Voice Disorders; RRP
Keywords: KTP; Blue light laser; laryngology; in office procedures
MeSH Terms: conditions — Voice Disorders | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Once consented, study participants will be randomized in a 1:1 ratio to one of two arms using a concealed permutated block randomization scheme to one of 2 arms - an experimental arm of BL laser treatment or a control arm of KTP laser treatment. Randomization sequence will be generated using a random number generator with randomly varying block sizes by the study statistician prior to the initiation of the study. Only the statistician and the research coordinator, who are not involved in the care of the patients, will know the randomization codes for allocation concealment. The intervention, i.e. type of laser used for treating the vocal fold lesions, is impossible to blind. Therefore this study is open-labeled. To further minimize bias from the open-labeled design, outcome measures will be collected and assessed by a blinded outcome assessor.
Who Masked: Outcomes Assessor
Masking Description: Only the statistician and the research coordinator, who are not involved in the care of the patients, will know the randomization codes for allocation concealment. To further minimize bias from the open-labeled design, outcome measures will be collected and assessed by a blinded outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KTP laser treatment (Active Comparator): All participants will complete a paper Voice Handicap Index-10 (VHI-10) questionnaire and laryngeal stroboscopy examination at baseline. Local anesthesia will be administered as per standard of care for in-office laryngeal procedures. KTP laser will be utilized to ablate the lesion of interest. Immediately following the procedure, participants will complete a VAS pain scale on paper. Participants will be asked to exercise 3 days of absolute voice rest following the procedure. All patients will have follow-up clinic appointments on POD 7, POD 30, and POD 90 after surgery. At each of the follow-up visit, the patients will fill out a paper VHI-10 questionnaire and undergo stroboscopic examination to assess vocal fold vibratory properties and closure, as well as residual lesions. During the first week post procedure, the participants will continue to complete a daily VAS at home for pain assessment.
  Interventions: Procedure: Laser treatment
- BL laser treatment (Experimental): The only difference in study procedures between the experimental arm and the control arm is that the experimental arm will use the BL laser. The post-operative instructions and follow-up schedule are identical.
  Interventions: Procedure: Laser treatment

INTERVENTIONS:
Procedure: Laser treatment — A flexible laser fiber will be utilized via a channelled laryngoscope to ablate the benign laryngeal lesions as per standard of care.

SUMMARY:
Preliminary investigations suggest that a novel blue light (BL) laser with a wavelength of 445nm is comparable to the commonly utilized KTP laser (532nm) for treatment of laryngeal pathologies. An animal study by the Principal Investigators showed that the blue light laser results in significantly less vocal fold scarring compared to the KTP laser, suggesting that the blue light laser may be a better instrument for treating vocal fold disease. However, there are no clinical studies directly comparing the two lasers on treatment of vocal fold pathology. The goal of the proposed study is to directly compare treatment outcomes of the BL laser and KTP laser for benign vocal fold lesions. All laser treatments will be performed in the office under local anesthesia as per standard of care. Outcome variables of interest will be compared between groups, including Voice Handicap Index-10 (VHI-10) score (measured at baseline, 1 week, 1 month, and 3 months post procedure), laryngeal stroboscopic findings (1 and 3 months post procedure), and intra-operative pain. This study will provide support that the blue light laser is a comparable alternative to the KTP laser and allow the addition of this novel laser to the armamentarium for treating vocal fold diseases.

DETAILED DESCRIPTION:
A novel blue light (BL) laser, TruBlue surgical laser, has recently been approved by Health Canada for use in the larynx. It has a wavelength of 445nm, which is within the same visible light spectrum as the KTP laser (532nm). It is a photoangiolytic laser like the KTP and can be delivered through a flexible fiber and therefore allowing the procedure to be performed in clinic under local anesthesia. Other advantages include better tissue cutting and increased portability. No clinical studies in the literature have directly compared the BL laser and KTP laser in the treatment of benign vocal fold lesions. The main objective of this proposal is to compare between-group differences in patient perception of voice handicap between BL laser and KTP laser for treatment of benign vocal fold lesions at 3 months compared to baseline. Given the PIs' previous work comparing vocal fold scarring induced by these two lasers in a rat model, we hypothesize that the blue light laser will be equally effective at treating benign vocal fold lesions as the KTP laser, resulting in improved VHI-10 score at 3 months post laser treatment compared to baseline.

The KTP laser has been a workhorse laser used in Otolaryngology/Laryngology for awake treatments of vocal fold lesions. However, it is phasing out of the market as the laser itself as well as the laser fibers compatible with this laser are no longer being manufactured. Therefore, Laryngologists are eagerly looking for an alternative to the KTP laser in order to fill this gap in care. The BL laser is cheaper in costs and more portable compared to the KTP. It also has better tissue cutting abilities which can be useful in treating certain vocal fold lesions such as vocal fold cancer and subglottic stenosis. This study is the first to directly compare treatment outcomes between the BL laser and KTP laser for vocal fold lesions. If the BL laser is shown to be comparable to the KTP in this clinical study, it lends support that this novel laser is indeed an excellent alternative to the KTP laser and can therefore be incorporated into routine patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Male and female, aged ≥ 18 years; and
4. Diagnosed with benign vocal fold lesions such as papillomas and polyps and who are candidates for elective in office laser treatment for these lesions.

Exclusion Criteria:

1. < 18 years old;
2. Current smokers;
3. Vocal fold lesions such as vocal fold leukoplakia and vocal fold cancer;
4. Systemic steroid use; and
5. History of systemic illness that can affect wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index-10 (VHI-10) | Change in VHI-10 score at 3 months
  VHI-10 is a validated 10-item questionnaire that quantifies the impact of voice limitations on the individual's overall daily function. It has a Cronbach's alpha of 0.90, indicating high internal consistency. It ranges from a score of 0 to 40. The higher the score, the worse the patient's perception of voice handicap. A score of ≥11 is abnormal. It is a standard of care at the Laryngology outpatient clinic at St. Michael's Hospital for patients to fill out the VHI-10 on paper independently before each clinic visit.

SECONDARY OUTCOMES:
Laryngeal stroboscopy | 3 months post op compared with baseline
  Laryngeal stroboscopy is controlled light illumination of the vocal folds during phonation timed to the frequency of the patient's voice. Images acquired during these flashes provide a slow motion-like view of vocal fold vibration during sound production to allow examination of vocal fold vibration and closure. Vocal fold mucosal vibration and closure pattern have been shown to be reliable and valid parameters to assess vocal fold healing after surgery of the vocal folds. These parameters will be collected as per standard of care at baseline, POD 7, POD 30, and POD 90 and will be judged by a blinded assessor (i.e. participant's non-treating Laryngologist who is not involved in his/her care) from video capture.
VAS pain scale | Immediately following laser treatment and daily for 1 week after the treatment
  A Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic which ranges across a continuum of values and cannot easily be directly measured. It will be ranked from a continuum scale of 1 to 10.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zeitels SM, Akst LM, Burns JA, Hillman RE, Broadhurst MS, Anderson RR. Office-based 532-nm pulsed KTP laser treatment of glottal papillomatosis and dysplasia. Ann Otol Rhinol Laryngol. 2006 Sep;115(9):679-85. doi: 10.1177/000348940611500905. PMID 17044539
- [Result] Hess MM, Fleischer S, Ernstberger M. New 445 nm blue laser for laryngeal surgery combines photoangiolytic and cutting properties. Eur Arch Otorhinolaryngol. 2018 Jun;275(6):1557-1567. doi: 10.1007/s00405-018-4974-8. Epub 2018 Apr 19. PMID 29675755
- [Result] Lin RJ, Iakovlev V, Streutker C, Lee D, Al-Ali M, Anderson J. Blue Light Laser Results in Less Vocal Fold Scarring Compared to KTP Laser in Normal Rat Vocal Folds. Laryngoscope. 2021 Apr;131(4):853-858. doi: 10.1002/lary.28892. Epub 2020 Aug 4. PMID 32750168